CLINICAL TRIAL: NCT03351699
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-4250 Monotherapy in Anti-Retroviral Therapy (ART)-Naive, HIV-1 Infected Subjects
Brief Title: Single-Dose Study of MK-4250 Monotherapy in Anti-Retroviral Therapy-Naive, Human Immunodeficiency Virus (HIV)-1 Infected Participants (MK-4250-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4250-002; 2017-001784-21 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Panel A: MK-4250 150 mg (Experimental): Participants will receive MK-4250 150 mg tablet by mouth on Day 1 after an 8-hour fast.
  Interventions: Drug: MK-4250
- Panel B: MK-4250 600 mg (Experimental): Participants will receive MK-4250 600 mg tablet by mouth on Day 1 after an 8-hour fast. The decision to enroll Panel B and the dose selected (i.e., ≤600 mg) will be made based on evaluation of pharmacokinetics and 7-day safety and viral load data from Panel A.
  Interventions: Drug: MK-4250
- Panel D: MK-4250 900 mg (Experimental): Participants will receive MK-4250 900 mg tablet by mouth on Day 1 after an 8-hour fast. The decision to enroll Panel D will be made upon completion of Panels A and B and evaluation of safety and viral load data from those panels.
  Interventions: Drug: MK-4250
- Panel E: MK-4250 ≤900 mg with a Low-fat Meal (Experimental): Participants will receive MK-4250 ≤900 mg tablet by mouth on Day 1 with a low-fat meal. The decision to enroll Panel E will be made upon completion of Panel D and evaluation of safety and viral load data from that panel.
  Interventions: Drug: MK-4250
- Panel F: MK-4250 ≤900 mg with a Moderate-fat Meal (Experimental): Participants will receive MK-4250 ≤900 mg tablet by mouth on Day 1 with a moderate-fat meal. The decision to enroll Panel F will be made upon completion of Panel D and evaluation of safety and viral load data from that panel. The decision to enroll Panel F will be made based on evaluation of PK and safety data from other studies with MK-4250.
  Interventions: Drug: MK-4250

INTERVENTIONS:
Drug: MK-4250 — MK-4250 tablets for oral administration

SUMMARY:
The study will evaluate the safety, tolerability, pharmacokinetics, and anti-retroviral activity of MK-4250 monotherapy in anti-retroviral therapy (ART)-naïve, HIV-1 infected participants. The primary hypothesis of the study is that at a dose that is sufficiently safe and generally well tolerated, MK-4250 has superior antiretroviral activity compared to a historical placebo, as measured by change from baseline in plasma HIV-1 ribonucleic acid (RNA) (log10 copies/mL) at 168 hours postdose.

DETAILED DESCRIPTION:
The study consists of 5 panels; Panel C (MK-4250 ≤600 mg) was removed from the study with Protocol Amendment 1.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-breast feeding female
* If female with reproductive potential: must demonstrate a serum β-human chorionic gonadotropin (β -hCG) level consistent with the nongravid state and agree to use a highly effective method of birth control until 30 days after the dose of trial drug
* If postmenopausal female: without menses for at least 1 year and has a documented follicle stimulating hormone (FSH) level in the postmenopausal range at pretrial (screening), AND/OR status post hysterectomy or oophorectomy
* Documented HIV-1 positive as determined by a positive Enzyme-linked Immunosorbent Assay (ELISA) or Quantitative Polymerase Chain Reaction (QT-PCR) with confirmation (e.g., Western Blot).
* No evidence at screening for mutations (e.g., E92Q, N55H, Q148K, Q148R and Y143R) affecting susceptibility to Integrase Strand Transfer Inhibitors (InSTIs)
* Diagnosed with HIV-1 infection ≥ 3 months prior to screening or confirmed chronic HIV infection
* Screening plasma Cluster of Differentiation (CD) 4+ T cell count of >200/mm^3
* Screening plasma HIV-1 RNA ≥5,000 copies/mL within 30 days prior to the treatment phase of this study
* Anti-retroviral therapy (ART)-naïve, which is defined as having never received any antiretroviral agent OR ≤30 consecutive days of an investigational antiretroviral agent which is not an InSTI and no exposure to such an investigational antiretroviral agent within 60 days prior to screening OR ≤60 consecutive days of combination ART which does not include an InSTI and no exposure to such ART within 60 days prior to screening
* Never received any InSTI
* Willing to receive no other ART for the duration of the treatment phase of this study
* Body Mass Index (BMI) ≤35 kg/m^2
* Other than HIV infection, have baseline health judged to be stable

Exclusion Criteria:

* Mentally or legally institutionalized / incapacitated, or significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder within the last 5 years
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, genitourinary or major neurological abnormalities or diseases
* History of cancer (malignancy). Exceptions: (1) adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix; (2) other malignancies which have been successfully treated ≥10 years prior to the pretrial (screening) visit with no evidence of recurrence; or, (3) deemed highly unlikely to sustain a recurrence for the duration of the trial
* History of significant multiple and/or severe allergies (e.g., food, drug, latex allergy); anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or non-prescription drugs or food; or hereditary galactose intolerance, lactose deficiency, or glucose-galactose malabsorption.
* Positive for hepatitis B surface antigen
* History of chronic hepatitis C (HCV) infection. Participants with a documented cure and/or a positive serologic test for HCV with a negative HCV viral load may be included
* Major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit
* Participated in another investigational trial within 4 weeks prior to the Day 1 dosing visit. The 4 week window will be derived from the date of the last trial medication and / or blood collection in a previous trial and/or an adverse event related to trial drug to the Day 1 dosing visit of the current trial
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of trial drug, throughout the trial, until the post-trial visit
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day. Participants who consume 4 glasses of alcoholic beverages per day may be enrolled
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day
* Excessive smoker (i.e., more than 10 cigarettes/day) and is unwilling to restrict smoking to ≤10 cigarettes per day
* Cardiac QTc interval ≥470 msec (for males) or ≥480 msec (for females)
* Positive urine drug screen (except for cannabis) at screening and/or predose; rechecks are allowed
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Charite Research Organisation GmbH ( Site 0001), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel A: MK-4250 150 mg: Participants received MK-4250 150 mg dose by mouth on Day 1 after an 8-hour fast.
- Panel B: MK-4250 600 mg: Participants received MK-4250 600 mg dose by mouth on Day 1 after an 8-hour fast. The decision to enroll Panel B and the dose selected (i.e., ≤600 mg) was made based on evaluation of pharmacokinetics and 7-day safety and viral load data from Panel A.
- Panel D: MK-4250 900 mg: Participants received MK-4250 900 mg dose by mouth on Day 1 after an 8-hour fast. The decision to enroll Panel D was made upon completion of Panels A and B and evaluation of safety and viral load data from those panels.
- Panel E: MK-4250 ≤900 mg With a Low-fat Meal: Participants received MK-4250 900 mg dose by mouth on Day 1 with a low-fat meal. The decision to enroll Panel E was made upon completion of Panel D and evaluation of safety and viral load data from that panel.
- Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal: Participants were to receive MK-4250 900 mg dose by mouth on Day 1 with a moderate-fat meal. The decision was made not to enroll Panel F because the scientific objectives were met following completion of Panel E.
Period: Overall Study
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Started | 6 | 6 | 6 | 6 | 0 (Panel F did not enroll, following evaluation of earlier Panel data.)
Completed | 6 | 6 | 6 | 6 | 0 (Panel F did not enroll, following evaluation of earlier Panel data.)
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Panel F did not enroll because the scientific objectives were met following completion of Panel E.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (8.1) | 32.5 (6.1) | 36.5 (8.9) | 35.5 (7.3) |  | 35.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 0 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 6 | 6 | 0 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 0 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Baseline Plasma HIV-1 Ribonucleic Acid (RNA) [Mean (Standard Deviation); unit: log10 copies/mL] — log10 HIV-1 RNA copies per mL of blood at baseline are presented.
  log10 copies/mL | 4.29394 (0.41200) | 4.42577 (0.39577) | 4.85677 (0.23790) | 4.42262 (0.37308) |  | 4.49978 (0.40099)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV-1 RNA Copies Per mL at 168 Hours
Description: Plasma HIV-1 RNA was measured at Baseline and 168 hours after dosing. The log10 plasma HIV-RNA copies/mL measurements from participants in each panel were pooled and analyzed based on a longitudinal data analysis model. The change from Baseline in plasma HIV-1 RNA in participants administered MK-4250 was compared with historical placebo data.
Time Frame: Baseline and Day 7
Population: All participants who complied with the protocol sufficiently to ensure data would likely exhibit the effects of treatment, according to the scientific model. Compliance included treatment exposure, measurement availability, and lack of major protocol deviations. Panel F did not enroll because the objectives were met following completion of Panel E.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies per mL
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
log10 copies per mL | -1.56 [-1.88 to -1.23] | -1.76 [-2.08 to -1.43] | -1.55 [-1.87 to -1.23] | -1.78 [-2.10 to -1.45] |
Statistical Analysis 1: Comparison: Panel A: MK-4250 150 mg; Test type: Superiority — Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a longitudinal data analysis (LDA) model containing fixed effects for study and time, and a random effect for participants. LS mean (95% confidence interval) for change from baseline at 168 hours post dose of pooled historical placebo was -0.03 log10 copies/mL (-0.14, 0.09); Posterior Mean Difference = -1.53 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-4250 and placebo at least 1.4 log10 copies/mL was 78%
Statistical Analysis 2: Comparison: Panel B: MK-4250 600 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -1.73 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-4250 and placebo at least 1.4 log10 copies/mL was 95%
Statistical Analysis 3: Comparison: Panel D: MK-4250 900 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -1.52 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-4250 and placebo at least 1.4 log10 copies/mL was 75%
Statistical Analysis 4: Comparison: Panel E: MK-4250 ≤900 mg With a Low-fat Meal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -1.75 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-4250 and placebo at least 1.4 log10 copies/mL was 96%

2. Primary Outcome: Percentage of Participants Experiencing ≥1 Adverse Events (AE)
Description: The percentage of participants experiencing ≥1 AE was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to Day 14
Population: Included all participants who received ≥1 dose of treatment. Panel F did not enroll because the scientific objectives were met following completion of Panel E.
Measure: Number; unit: Percentage of Participants
Groups:
- Screening: This arm is all participants from all treatment arms, analyzed during the period prior to receipt of any study intervention.
Arm/Group | Screening | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 0
Percentage of Participants | 8.3 | 83.3 | 66.7 | 83.3 | 66.7 |

3. Primary Outcome: Percentage of Participants Who Discontinued Study Due to an Adverse Event (AE)
Description: The percentage of participants who discontinued from the study due to an adverse event was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Screening | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 0
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 |

4. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to Last Measurable Concentration (AUC0-last) for MK-4250
Description: The area under the concentration-time curve up to the last measurable concentration (AUC0-last) of MK-4250 in plasma was calculated.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 120, 168, 192, and 240 hours after administration of MK-4250. For Panel B only, the first three participants additionally had a 72-hour postdose time, and no 240-hour postdose time.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hour
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
μM·hour | 774 (54) | 2040 (17.1) | 2390 (35) | 3860 (44.3) |

5. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to Infinity (AUC0-inf) for MK-4250
Description: The area under the concentration-time curve extrapolated to infinity (AUC0-inf) of MK-4250 in plasma was calculated.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hour
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
μM·hour | 785 (54.6) | 2120 (18.4) | 2450 (35.9) | 4010 (47.6) |

6. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 168 Hours (AUC0-168) for MK-4250
Description: The area under the concentration-time curve up to 168 hours (AUC0-168) of MK-4250 in plasma was calculated.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 120, and 168 hours after administration of MK-4250. For Panel B only, the first three participants additionally had a 72-hour postdose time.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·Hour
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
μM·Hour | 751 (52.6) | 1980 (16.7) | 2280 (34.1) | 3640 (41.2) |

7. Secondary Outcome: Maximum Concentration (Cmax) of MK-4250 Reached in Plasma
Description: The maximum concentration (Cmax) of MK-4250 in plasma was observed.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
μM | 16.6 (46.7) | 37.6 (26) | 43.5 (32.7) | 65 (25.8) |

8. Secondary Outcome: Concentration of MK-4250 at 168 Hours (C168hr)
Description: The concentration of MK-4250 at 168 hours postdose (C168hr) was observed.
Time Frame: 168 hours after administration of MK-4250.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
μM | 0.558 (117) | 2.2 (57.4) | 2.38 (63.8) | 4.37 (96.4) |

9. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-4250
Description: The apparent terminal half-life (t1/2) of MK-4250 in plasma was calculated.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
Hours | 35.9 (22.9) | 38.5 (31.9) | 44.1 (17.1) | 48.4 (32.1) |

10. Secondary Outcome: Apparent Clearance (CL/F) of MK-4250
Description: The apparent clearance (CL/F) of MK-4250 in plasma was calculated.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/Hour
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
Liters/Hour | 0.456 (54.6) | 0.676 (18.4) | 0.879 (35.9) | 0.536 (47.6) |

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of MK-4250
Description: The apparent volume of distribution (Vz/F) of MK-4250 in plasma was calculated.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
Liters | 23.6 (45.1) | 37.6 (23.5) | 56 (31.7) | 37.4 (17.5) |

12. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-4250 Reached in Plasma
Description: The time to maximum concentration (Vz/F) of MK-4250 in plasma was calculated.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A: MK-4250 150 mg | Panel B: MK-4250 600 mg | Panel D: MK-4250 900 mg | Panel E: MK-4250 ≤900 mg With a Low-fat Meal | Panel F: MK-4250 ≤900 mg With a Moderate-fat Meal
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
Hours | 4.00 [1.00 to 4.00] | 4.00 [4.00 to 6.00] | 4.00 [4.00 to 6.00] | 4.00 [4.00 to 8.00] |

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Groups:
- Screening: This group represents all participants during their individual screening phase, approximately 4 weeks prior to first dose. No intervention was provided during this time.
- Panel A: 150 mg MK-4250: Participants received MK-4250 150 mg tablet by mouth on Day 1 after an 8-hour fast.
- Panel B: 600 mg MK-4250: Participants received MK-4250 600 mg tablet by mouth on Day 1 after an 8-hour fast. The decision to enroll Panel B and the dose selected (i.e., ≤600 mg) was made based on evaluation of pharmacokinetics and 7-day safety and viral load data from Panel A.
- Panel D: 900 mg MK-4250: Participants received MK-4250 900 mg tablet by mouth on Day 1 after an 8-hour fast. The decision to enroll Panel D was made upon completion of Panels A and B and evaluation of safety and viral load data from those panels.
- Panel E: 900 mg MK-4250, With a Low Fat Meal: Participants received MK-4250 ≤900 mg tablet by mouth on Day 1 with a low-fat meal. The decision to enroll Panel E was made upon completion of Panel D and evaluation of safety and viral load data from that panel.
Arm/Group | Screening | Panel A: 150 mg MK-4250 | Panel B: 600 mg MK-4250 | Panel D: 900 mg MK-4250 | Panel E: 900 mg MK-4250, With a Low Fat Meal
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/24 | 5/6 | 4/6 | 5/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening (N=24) | Panel A: 150 mg MK-4250 (N=6) | Panel B: 600 mg MK-4250 (N=6) | Panel D: 900 mg MK-4250 (N=6) | Panel E: 900 mg MK-4250, With a Low Fat Meal (N=6)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication (or after public disclosure of the results at www.clinicaltrials.gov if multicenter manuscript is not planned), an investigator and colleagues may publish their data independently. Sponsor must have opportunity to review proposed abstracts, manuscripts or presentations 45 days prior to submission for publication/presentation. Confidential information must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT03351699/Prot_SAP_000.pdf